CLINICAL TRIAL: NCT05014919
Title: A Double-blind, Randomized, Placebo-controlled, Multicentre, Relapse-prevention Study of Vortioxetine in Paediatric Patients Aged 7 to 11 Years With Major Depressive Disorder
Brief Title: Vortioxetine to Prevent Return of Symptoms in Children With Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated based on new efficacy data from another study.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13546A; 2010-020493-42 (EudraCT Number)
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vortioxetine -open label treatment period (Experimental): Vortioxetine - 5, 10, 15, and 20 mg/day, film-coated tablets, orally once daily.
  Patients will receive a targeted dose of 10 mg/day vortioxetine, however the investigator has the possibility to adjust the dose in case of unsatisfactory response or in case of dose-limiting adverse events.
  Interventions: Drug: Vortioxetine
- Vortioxetine -double-blind relapse prevention period (Experimental): Vortioxetine - 5, 10, 15, and 20 mg/day, encapsulated film-coated tables, orally once daily.
  In the double-blind period, the patients will continue on the same fixed dose as during the end of the open label period
  Interventions: Drug: Vortioxetine
- Placebo -double-blind relapse prevention period (Placebo Comparator): Placebo - encapsulated tablets, orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Tablets
  Other Names: Brintellix; Trintellix
  Arms: Vortioxetine -double-blind relapse prevention period; Vortioxetine -open label treatment period
Drug: Placebo — Tablets
  Arms: Placebo -double-blind relapse prevention period

SUMMARY:
The purpose of this study is to find out if vortioxetine is better than placebo (sugar pills) in preventing depression in children who improved when treated with vortioxetine.

DETAILED DESCRIPTION:
The study consists of a 12-week open-label, flexible-dose treatment period with vortioxetine, followed by a 26-week, randomized, double-blind, fixed-dose, placebo-controlled relapse-prevention period. There will be a safety follow up 4 weeks after the end of the 26-week double-blind treatment period.

The study population will include 'de novo' participants as well as 'rollover' participants from other paediatric vortioxetine studies 12709A (NCT02709655) and 12712A (NCT02871297), who, in the investigator's opinion, could benefit from continued treatment with vortioxetine.

ELIGIBILITY:
Inclusion Criteria:

De novo participants

* The participant has a primary diagnosis of MDD according to DSM-5™ although co-morbid anxiety disorders will be permitted (except Post Traumatic Stress Disorder (PTSD) and Obsessive Compulsive Disorder (OCD)).
* The participant has a CDRS-R total score ≥45 at the Screening and Baseline Visits.
* The participant has a Clinical Global Impression - Severity of Illness (CGI-S) ≥4 at the Screening and Baseline Visit

Exclusion Criteria:

* The participant receives ongoing current psychotherapy that is planned to be intensified. Interpersonal psychotherapy (IPT) or cognitive behavioural therapy (CBT) are not allowed.
* The participant presents with, or has a history of, an Axis I (DSM-5TM) diagnosis of Bipolar Disorder, PTSD, OCD, Autism, Pervasive Developmental Disorder (PDD), or Schizophrenia or Schizoaffective Disorder.
* The participant has a diagnosis of attention-deficit/hyperactivity disorder (ADHD) and is not maintained on a stable dose of a methylphenidate or amphetamine for a minimum of 4 weeks prior to the study treatment.
* The participant has attempted suicide or is at significant risk of suicide

Other inclusion and exclusion criteria may apply.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (17):
- United States (3):
  - Alliance for Research, Long Beach, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - AIM Trials, LLC, Plano, Texas
- Colombia (3):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA LTDA IPS., Barranquilla, Atlántico
  - Centro de investigaciones del Sistema Nervioso SAS Grupo CISNE SAS, Bogotá, DC
  - Psynapsis Salud Mental S.A., Pereira, Risaralda Department
- Linda Keruze's Psychiatric Center, LLC, Liepāja, Latvia
- Mexico (3):
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - BIND Investigaciones S.C, San Luis Potosí City, San Luis Potosí
  - SINACOR - Centro para el Desarrollo de la Medicina Y De Asistencia Medica Especializada S.C, Culiacan de Rosales, Sinaloa
- Poland (2):
  - Przychodnia Syntonia Izabela Chojnowska-Cwiakala, Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska, Poznan
- Russia (4):
  - Medicorehabilitation Research Center Phoenix, Rostov-on-Don, Rostov State
  - GUZ Engels Psychiatric Hospital, Engel's
  - Rostov State Medical University of the Minzdravsotsrazvitiya of Russia, Rostov-on-Don
  - Nebbiolo LLC, Tomsk
- Odessa Regional Psychiatry Hospital No. 2, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included de novo participants as well as rollover participants from other paediatric vortioxetine studies (Studies 12709A [NCT02709655] and 12712A [NCT02871297]) who, in the investigator's opinion, would benefit from continued treatment with vortioxetine.
Pre-assignment Details: Rollover participants from Study 12709A enrolled to the open-label period and rollover participants (remitters) from Study 12712A randomized to the double-blind period. Overall, 35 participants were treated in this study: 33 participants in the open-label period (24 de novo participants and 9 rollover participants from Study 12709A) and 4 participants in the double-blind period (2 of whom rolled-over from Study 12712A).
Groups:
- Open-Label Treatment: Vortioxetine: Participants initiated treatment with vortioxetine tablets 5 milligrams (mg)/day orally for the first 2 days and thereafter they received 10 mg/day vortioxetine. Based on the response and dose-limiting adverse events (AEs), vortioxetine dose could be up- or down-titrated with 5 mg/day to a maximum of 20 mg/day during the first 8 weeks. From Week 8 to Week 12, the dose remained fixed.
- Double-Blind Relapse Prevention: Vortioxetine: Participants continued on the same fixed dose of vortioxetine as during the end of the open-label period for 26 weeks in the double-blind relapse prevention period.
- Double-Blind Relapse Prevention: Placebo: Participants received placebo for 26 weeks in the double-blind relapse prevention period.
Period: Open-Label (12 Weeks)
Arm/Group | Open-Label Treatment: Vortioxetine | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Started | 33 (24 de novo and 9 rollover participants) | 0 | 0
Received at Least 1 Dose of Study Drug | 33 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 28 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Based on Sponsor Information of Results From Vortioxetine Study | 15 | 0 | 0
Not completed — Sponsor Decision | 4 | 0 | 0
Not completed — Study Terminated by Sponsor | 5 | 0 | 0
Period: Double-Blind (26 Weeks)
Arm/Group | Open-Label Treatment: Vortioxetine | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Started | 0 | 2 (1 from open-label period and 1 from study 12712A) | 2 (1 from open-label period and 1 from study 12712A)
Received at Least 1 Dose of Study Drug | 0 | 2 | 2
Completed | 0 | 1 | 0
Not Completed | 0 | 1 | 2
Not completed — Study Terminated by Sponsor | 0 | 0 | 1
Not completed — Based on Sponsor Information of Results From Vortioxetine Study | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All-patients-enrolled (APES): all participants enrolled to the 12-week open-label treatment period who took at least 1 dose of study drug. Full analysis set (FAS): all participants randomized to the 26-week double-blind treatment period who took at least 1 dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-Label Treatment: Vortioxetine | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo | Total
Number analyzed (Participants) | 33 | 2 | 2 | 37
Age, Customized [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind arms.
  Participants
    Open-Label Treatment: number analyzed (Participants) | 33 | 0 | 0 | 33
    Open-Label Treatment: Children (2-11 years) | 27 | 0 | 0 | 27
    Open-Label Treatment: Adolescents (12-17 years) | 6 | 0 | 0 | 6
    Double-Blind Relapse Prevention: number analyzed (Participants) | 0 | 2 | 2 | 4
    Double-Blind Relapse Prevention: Children (2-11 years) | 0 | 2 | 2 | 4
    Double-Blind Relapse Prevention: Adolescents (12-17 years) | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind arms.
  Participants
    Open-Label Treatment: number analyzed (Participants) | 33 | 0 | 0 | 33
    Open-Label Treatment: Female | 18 | 0 | 0 | 18
    Open-Label Treatment: Male | 15 | 0 | 0 | 15
    Double-Blind Relapse Prevention: number analyzed (Participants) | 0 | 2 | 2 | 4
    Double-Blind Relapse Prevention: Female | 0 | 1 | 1 | 2
    Double-Blind Relapse Prevention: Male | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind arms.
  Participants
    Open-Label Treatment: number analyzed (Participants) | 33 | 0 | 0 | 33
    Open-Label Treatment: Hispanic or Latino | 18 | 0 | 0 | 18
    Open-Label Treatment: Not Hispanic or Latino | 15 | 0 | 0 | 15
    Open-Label Treatment: Unknown or Not Reported | 0 | 0 | 0 | 0
    Double-Blind Relapse Prevention: number analyzed (Participants) | 0 | 2 | 2 | 4
    Double-Blind Relapse Prevention: Hispanic or Latino | 0 | 2 | 1 | 3
    Double-Blind Relapse Prevention: Not Hispanic or Latino | 0 | 0 | 0 | 0
    Double-Blind Relapse Prevention: Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data are being reported separately for the open-label and double-blind arms.
  Participants
    Open-Label Treatment: number analyzed (Participants) | 33 | 0 | 0 | 33
    Open-Label Treatment: White | 13 | 0 | 0 | 13
    Open-Label Treatment: Black or African American | 3 | 0 | 0 | 3
    Open-Label Treatment: Asian | 1 | 0 | 0 | 1
    Open-Label Treatment: Other | 16 | 0 | 0 | 16
    Double-Blind Relapse Prevention: number analyzed (Participants) | 0 | 2 | 2 | 4
    Double-Blind Relapse Prevention: White | 0 | 0 | 2 | 2
    Double-Blind Relapse Prevention: Black or African American | 0 | 0 | 0 | 0
    Double-Blind Relapse Prevention: Asian | 0 | 0 | 0 | 0
    Double-Blind Relapse Prevention: Other | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse in the Double-blind Period
Description: Relapse was defined as either a total score ≥40 on the Children Depression Rating Scale Revised Version (CDRS-R) with a history of 2 weeks of clinical deterioration, or clinical deterioration as judged by the clinician. The CDRS-R is rated by a clinician following interviews with the child and parent and consists of 17 items out of which 3 items rate nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items are rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) are scored on a 5-point scale from 1 to 5. A rating of 1 indicates normal functioning and a higher number indicates a greater degree of depression. The total score ranges from 17 (normal) to 113 (severe depression).
Time Frame: From randomization to Week 26 in the double-blind treatment period
Population: Due to the early termination of study and limited number of participants who completed the double-blind period, the efficacy analyses were not performed and data were not collected for this outcome measure.
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Relapse Rate in the Double-blind Period: Percentage of Participants With Relapse
Description: Relapse was defined as either a total score ≥40 on the CDRS-R with a history of 2 weeks of clinical deterioration, or clinical deterioration as judged by the clinician. The CDRS-R is rated by a clinician following interviews with the child and parent and consists of 17 items out of which 3 items rate nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items are rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) are scored on a 5-point scale from 1 to 5. A rating of 1 indicates normal functioning and a higher number indicates a greater degree of depression. The total score ranges from 17 (normal) to 113 (severe depression).
Time Frame: From randomization to Week 26 in the double-blind treatment period
Population: as for outcome 1
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale - Revised Version (CDRS-R) Total Score at Week 26
Description: The CDRS-R is a clinician-rated scale to measure the severity of depression in children and adolescents. The CDRS-R is rated by a clinician following interviews with the child and parent and consists of 17 items out of which 3 items rate nonverbal observations (listless speech, hypoactivity, and depressed affect). Fourteen items are rated on a 7-point scale from 1 to 7, and 3 items (sleep disturbance, appetite disturbance, and listless speech) are scored on a 5-point scale from 1 to 5. A rating of 1 indicates normal functioning and a higher number indicates a greater degree of depression. The total score ranges from 17 (normal) to 113 (severe depression).
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Score at Week 26
Description: The CGI-S provides the clinician's impression of the participant's current state of mental illness. The clinician uses his or her clinical experience of this participant population to rate the severity of the participant's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Score at Week 26
Description: The CGI-I provides the clinician's impression of the participant's improvement (or worsening). The clinician assesses the participant's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 26
Population: as for outcome 1
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Paediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Total Score (Items 1 to 14) at Week 26
Description: The PQ-LES-Q is a participant-rated scale designed to assess satisfaction with life. It is an adaptation of the Quality of Life Enjoyment and Satisfaction Questionnaire, which is used to measure quality of life in adults. The PQ-LES-Q consist of 15 items, item 1 to 14 assess the degree of satisfaction experienced by participants in various areas of daily functioning, and item 15 allows participants to summarise their experience in a global rating. Each item is rated on a 5-point scale from 1 (very poor) to 5 (very good). The total score range of item 1 to 14 is 14 to 70, with higher scores indicating greater satisfaction.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Plasma Concentration of Vortioxetine
Time Frame: From randomization to Week 26 in the double-blind treatment period
Population: Due to early termination of the study, the pharmacokinetic analyses were not performed and the data were not collected.
Arm/Group | Double-Blind Relapse Prevention: Vortioxetine | Double-Blind Relapse Prevention: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) up to Week 42
Description: All-patients-enrolled (APES) included all participants enrolled to the 12-week open-label, flexible-dose treatment period who took at least 1 dose of study drug. All-patients-randomized set (APRS) included all participants randomized to the 26-week double-blind treatment period.
Groups:
- Open-Label Treatment: Vortioxetine: Participants initiated treatment with vortioxetine tablets 5 mg/day orally for the first 2 days and thereafter they received 10 mg/day vortioxetine. Based on the response and dose-limiting AEs, vortioxetine dose could be up- or down-titrated with 5 mg/day to a maximum of 20 mg/day during the first 8 weeks. From Week 8 to Week 12, the dose remained fixed.
Arm/Group | Open-Label Treatment: Vortioxetine | Double-Blind Relapse Prevention: Placebo | Double-Blind Relapse Prevention: Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 8/33 | 1/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment: Vortioxetine (N=33) | Double-Blind Relapse Prevention: Placebo (N=2) | Double-Blind Relapse Prevention: Vortioxetine (N=2)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on new efficacy data from another study. The main primary and secondary efficacy objectives were not assessed due to termination of the study and the limited number of participants who completed the double-blind period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT05014919/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT05014919/SAP_003.pdf